CLINICAL TRIAL: NCT01848288
Title: Intra-Operative Metrics and Clinical Outcomes After Cataract Surgery With the CENTURION® Vision System and the INFINITI® Vision System
Brief Title: Intra-Operative Metrics With CENTURION® and INFINITI® Vision Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: M-13-006
Record Dates: First submitted 2013-05-01; First posted 2013-05-07 (Estimated); Results first posted 2015-03-09 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Cataract
Keywords: Cataract; Phacoemulsification; Cumulative Dissipated Energy (CDE)
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CENTURION (Experimental): First surgical eye randomized to CENTURION® Vision System, with second surgical eye (fellow eye) assigned to INFINITI® Vision System. Second eye surgery conducted within 14 days of the first eye surgery. Duration of surgery less than 30 minutes each eye.
  Interventions: Device: CENTURION® Vision System (CVS); Device: INFINITI® Vision System (IVS)
- INFINITI (Active Comparator): First surgical eye randomized to INFINITI® Vision System, with second surgical eye (fellow eye) assigned to CENTURION® Vision System. Second eye surgery conducted within 14 days of the first eye surgery. Duration of surgery less than 30 minutes each eye.
  Interventions: Device: CENTURION® Vision System (CVS); Device: INFINITI® Vision System (IVS)

INTERVENTIONS:
Device: CENTURION® Vision System (CVS) — Phacoemulsification aspiration platform, with configuration consisting of Centurion® Vision System Phaco Emulsifier Aspirator, 45° Balanced ultrasonic tip, and INTREPID Ultra Infusion Sleeve, for use during routine cataract extraction by phacoemulsification with intraocular lens implantation.
Device: INFINITI® Vision System (IVS) — Phacoemulsification aspiration platform, with configuration consisting of Infiniti® Vision System Phaco Emulsifier Aspirator, 45° Mini Flared Kelman tip, and Ultra Infusion Sleeve, for use during routine cataract extraction by phacoemulsification with intraocular lens implantation.

SUMMARY:
The purpose of this study is to evaluate intra-operative phacoemulsification machine metrics after phacoemulsification with the CENTURION® vision system configuration compared with the INFINITI® vision system configuration.

ELIGIBILITY:
Inclusion Criteria:

* Eligible to undergo cataract extraction via phacoemulsification with primary ACRYSOF Intraocular Lens (IOL) implantation;
* Free of severe disease(s)/condition(s) listed in the "Warnings" and "Precautions" section of implanted ACRYSOF IOL;
* Willing to undergo second eye surgery within 14 days of first eye surgery;
* Willing and able to understand/sign a written Informed Consent Document;
* Willing and able to return for scheduled follow-up examinations;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Planned multiple procedures at the time of surgery or during the course of the study (eg, LASIK, LRI, etc.);
* Previous intraocular or corneal surgery of any kind;
* Poorly dilating pupil;
* Severe retinal disorders (eg, macular degeneration, proliferative diabetic retinopathy);
* Corneal disease (eg, herpes simplex, herpes zoster, etc) or retinal detachment;
* Severe conditions that per Investigator's clinical judgment would increase the operative risk or confound the result of this investigation;
* Female patients who are pregnant, lactating, or planning to be pregnant during the course of the study;
* Currently participating in another drug or device clinical trial, or participated in another drug or device clinical trial within 30 days of enrollment into this trial;
* Other protocol-defined exclusion criteria may apply.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2013-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Hayes, MS, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 2 investigative sites located in the US and 1 investigative site located in Spain.
Pre-assignment Details: Of the 112 enrolled, 12 participants were exited as screen failures prior to randomization. One participant was randomized twice in error. This reporting group includes all randomized participants (100).
Groups:
- Overall: First surgical eye randomly assigned to CENTURION® Vision System or INFINITI® Vision System, with the second surgical eye (fellow eye) assigned to the alternative group.
Period: Overall Study
Arm/Group | Overall
Started | 100
Completed | 97 (Two subjects were discontinued prior to undergoing surgery.)
Not Completed | 3
Not completed — Death | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: This reporting group includes all participants randomized to a surgical system.
Arm/Group | Overall
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.0 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 33

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Dissipated Energy
Description: Cumulative Dissipated Energy (CDE) is an estimation of the energy at the incision site experienced during the removal of cataractous lens and is measured in %-secs. The incision is defined as 5.6mm back from the cutting edge of the tip. A lower CDE indicates that less energy was present at the incision site.
Time Frame: Day 0 (operative day), each eye
Population: This analysis population includes all participants who were randomized to a surgical system and had non-missing values at the specific time point for each arm group, respectively.
Measure: Least Squares Mean (Standard Error); unit: percent-seconds
Groups:
- CENTURION Vision System: CENTURION® Vision System randomly assigned to first surgical eye, with INFINITI® Vision System assigned to second surgical eye (fellow eye). Each eye received a single treatment with estimated duration of less than 30 minutes. The second eye surgery occurred within 14 days of first eye surgery.
- INFINITI Vision System: INFINITI® Vision System randomly assigned to first surgical eye, with CENTURION® Vision System assigned to second surgical eye (fellow eye). Each eye received a single treatment with estimated duration of less than 30 minutes. The second eye surgery occurred within 14 days of first eye surgery.
Arm/Group | CENTURION Vision System | INFINITI Vision System
Number analyzed (Participants) | 98 | 97
percent-seconds | 4.32 (0.28) | 7.11 (0.28)

2. Primary Outcome: Aspiration (ASP) Fluid Used
Description: Aspiration fluid used is the amount of aspiration fluid used during the removal of the cataractous lens. A lower value indicates that less fluid was removed from the eye.
Time Frame: Day 0 (operative day), each eye
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: grams
Arm/Group | CENTURION Vision System | INFINITI Vision System
Number analyzed (Participants) | 98 | 97
grams | 46.56 (1.39) | 52.68 (1.40)

3. Secondary Outcome: Aspiration Time
Description: Aspiration Time indicated the amount of time the system was aspirating during the removal of the cataractous lens. A lower value indicates that the surgeon spent less time aspirating fluid and material from the eye during surgery.
Time Frame: Day 0 (operative day), each eye
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | CENTURION Vision System | INFINITI Vision System
Number analyzed (Participants) | 98 | 97
seconds | 151.85 (4.08) | 167.63 (4.09)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (01 Jul 2013 - 07 Feb 2014). This analysis group includes all participants who were randomized and treated.
Description: An AE was defined as any untoward medical occurrence in a subject who is administered a clinical trial treatment (ie, implant with an investigational device) regardless of whether or not the event has a causal relationship with the treatment.
Groups:
- Overall: First surgical eye randomly assigned to CENTURION® Vision System or INFINITI® Vision System, with the second surgical eye (fellow eye) assigned to the alternative group. For non-ocular adverse events, "at risk" population is included with unit of "subjects." For ocular adverse events, "at risk" population is included with unit of "eyes by treatment group."
Arm/Group | Overall
Serious Adverse Events (participants affected / at risk) | 2/98
Other Adverse Events (participants affected / at risk) | 11/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall (N=98)
Myocardial infarction (Cardiac disorders) | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Overall (N=98)
Vitreous detachment (Centurion) (Eye disorders) | 6
Intraocular pressure increased (Centurion) (Investigations) | 4
Vitreous detachment (Infiniti) (Eye disorders) | 6
Intraocular pressure increased (Infiniti) (Investigations) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.